CLINICAL TRIAL: NCT00797953
Title: A Phase II, Double Blind, Placebo-controlled, Randominzed, Multi-Center, Parallel Group Study to Evaluate the Efficacy and Safety of T89 in Patient With Chronic Stable Angina Pectoris
Brief Title: Phase II Multi-Center Study of T89 to Treat Chronic Stable Angina
Acronym: T89 phase 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: T89-005-0003-US
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Angina Pectoris
Keywords: Angina Pectoris Treatment
MeSH Terms: conditions — Angina Pectoris | interventions — T89 herbal drug

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose (Experimental): 2 capsules of T89 with 1 placebo capsule each time, twice daily. The daily dose is 250 mg.
  Interventions: Drug: T89
- High dose (Experimental): 3 capsules of T89 each time, twice daily. The daily dose is 375 mg
  Interventions: Drug: T89
- Placebo (Placebo Comparator): 3 placebo capsules (PC) each time, twice per day. The daily dose is 0 mg.
  Interventions: Drug: T89

INTERVENTIONS:
Drug: T89 — A two-herb botanical drug product in 62.5mg capsule formulation. It is to be used as 125mg or 187.5mg twice daily.
  Other Names: Dantonic Capsule; Cardiotonic Pills

SUMMARY:
The purpose of this study is to determine the anti-angina effect and dose response of T89, a 2-herb botanical drug product, in patients with chronic stable angina pectoris in the United States.

DETAILED DESCRIPTION:
T89 is a modernized and industrialized version of a traditional Chinese herbal medicine. T89 was approved for marketing as a drug, for the treatment of chronic stable angina pectoris due to coronary heart disease, by the State Food and Drug Administration (SFDA) of China in 1993. There were more than 2 billion doses have been prescribed or used, in about 10,000,000 subjects, in short or long-term administration worldwide.

The product is also marketed, as a drug, in Russia, South Korea, Mongolia, Singapore, Vietnam, and South Africa. The current study is to determine the anti-angina effect and dose response of T89 in patients with chronic stable angina pectoris in the United States.

T89 consists of Danshen (Radix Salviae Miltiorrhizae, RSM) and Sanqi (Radix Notoginseng, RN) as active constitutes, and using Borneol as transporting enhancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be between the ages of 18 and 80 years.
2. Females of childbearing potential must have a negative pregnancy test, not be breast feeding and established on a method of contraception that in the investigator's opinion is acceptable. Females must agree to remain on their established method of contraception through their participation in the study.
3. Evidence of coronary artery disease that consists of a well-documented medical history (over 3 months prior to the enrollment) of myocardial infarction or significant coronary artery disease with noninvasive or angiographic confirmation.
4. Symptoms that support the diagnosis of chronic angina and/or a history of an abnormal exercise response limited by angina and/or electrocardiograph (ECG) changes.
5. Moderate angina pectoris (Class II or Class III, Grading of Angina Pectoris by the Canadian Cardiovascular Society Classification System)
6. Naive patient or patient who's Total Exercise Duration (TED) is between 3 to 7 minutes in ETT on Standard Bruce Protocol, and the difference in TED must be no more than 15% between the two screen examinations on day -7 and day 0
7. All anti-angina regimen (except short-acting nitroglycerin, and one beta-blocker or calcium channel blocker), warfarin or other oral anticoagulants which were used prior to this initial visit can be discontinued.
8. Patient must understand and be willing, able and likely to comply with all study procedures and restrictions and comprehends the verbal rating scales and diary cards.
9. Patient must be able to give voluntary written informed consent.

Exclusion Criteria:

1. With contraindication to perform treadmill Exercise Tolerance Test (ETT).
2. Pre-exercise ST-segment depression of at least 1 mm in any lead, left bundle branch block, digoxin therapy, Left Ventricular Hypertrophy (LVH) and Wolff-Parkinson-White (WPW) syndrome or other factors that could interfere with exercise electrocardiograph interpretation.
3. Clinically significant arrhythmias or atrioventricular conduction block greater than first degree.
4. Clinically significant co-morbidities, including hepatic or renal dysfunction, pulmonary hypertension, chronic obstructive pulmonary disease, history of cerebral hemorrhage, or seizure disorders that required anticonvulsant medication.
5. History of congestive heart failure, unstable angina, severe valvular disease, severe hypertension, severe anemia, suspected or known dissecting aneurysm, acute myocarditis or pericarditis, thrombophlebitis or pulmonary embolism or recent myocardial infarction within three months of study entry.
6. History of bleeding diathesis, or is on warfarin.
7. Implanted pacemaker.
8. Aspirin and/or statins started less than 14 days prior to the signing of informed consent.
9. Pregnancy or lactation.
10. Inability to discontinue existing chronic nitrate regimen (e.g. long acting nitroglycerin) and allow only short-acting nitroglycerin and one beta-blocker or calcium channel blocker.
11. Clinical trials/experimental medication:

    * Participation in any other clinical trial or receipt of an investigational drug within 90 days prior to initial visit.
    * Those patients unable, in the opinion of the investigator, to comply fully with the trial requirements.
    * Previous participation in this study.
12. Substance abuse. Patients with a recent history (within the last 2 years) of alcoholism or known drug dependence.
13. Patient is a family member or relative of the study site staff.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Total Exercise Duration (TED) change from screen baseline value in Exercise Tolerance Test (ETT) on Standard Bruce Protocol at trough drug levels at the end of the 4th and 8th week of treatment compared to placebo. | 12 weeks

SECONDARY OUTCOMES:
Frequency of weekly angina episodes | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jason Zhixin Guo, MD, Study Director — Tasly Pharmaceuticals Co. Ltd.
Locations (15):
- United States (15):
  - Paradigm Clinical, Inc., Tucson, Arizona
  - Robert M. Karns, A Medical Corporation, Beverly Hills, California
  - Inland Heart Doctors, Corona, California
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Great Lakes Research Group, Inc, Bay City, Michigan
  - Marc Kozinn Associates, Williamsville, New York
  - Oklahoma Cardiovascular & Hypertension, Oklahoma City, Oklahoma
  - Three Rivers Medical Associates, Columbia, South Carolina
  - East Texas Cardiology, Houston, Texas
  - Northwest Houston Cardiology, Houston, Texas
  - Northwest Heart Center, Tomball, Texas
  - National Clinical Research-Norfolk, Inc, Norfolk, Virginia
  - Gemini Scientific, LLC, Madison, Wisconsin

REFERENCES:
- See also: Manufacture — http://WWW.TASLY.COM